CLINICAL TRIAL: NCT01065246
Title: Phase II Open Label Study to Evaluate the Safety of a Second I.P. Infusion Cycle of Catumaxomab in Patients With Malignant Ascites Due to Carcinoma, Requiring Their First Therapeutic Puncture After Treatment in the CASIMAS Study
Brief Title: Safety Study of Second Intraperitoneal (I.P.) Infusion Cycle of Catumaxomab in Patients With Malignant Ascites
Acronym: SECIMAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neovii Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP-CAT-AC-04; 2009-014076-22 (EudraCT Number)
Record Dates: First submitted 2010-01-13; First posted 2010-02-09 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-08

CONDITIONS: Malignant Ascites Due to Epithelial Carcinoma
Keywords: malignant ascites; second cycle; trifunctional
MeSH Terms: interventions — catumaxomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- catumaxomab (Experimental)
  Interventions: Drug: catumaxomab

INTERVENTIONS:
Drug: catumaxomab — 4 intraperitoneal infusions within 11 days administered over 3 hours via an indwelling catheter at the following doses: 10 - 20 - 50 - 150 µg catumaxomab
  Other Names: Removab

SUMMARY:
This phase II single arm, open-label study investigate the safety of a second cycle of catumaxomab in patients with malignant ascites due to carcinoma, requiring their first therapeutic puncture after treatment in the CASIMAS study.

DETAILED DESCRIPTION:
Up to 30 evaluable patients from the CASIMAS study will be enrolled. Catumaxomab will be infused intraperitoneally with 3hour constant-rate infusions 4 times within 11 days with ascending dosages (10 - 20 - 50 - 150 µg).

ELIGIBILITY:
Inclusion Criteria:

* patients who have completed 4 infusions of catumaxomab in the CASIMAS study
* age >= 18 years
* Karnofsky index >= 60 %
* patients with malignant ascites requiring their first therapeutic ascites paracentesis after at least 60days following last catumaxomab infusion in the CASIMAS study
* Patients where standard therapy is either not available or no longer feasible

Exclusion Criteria:

* acute or chronic infection
* concomitant treatment with investigational products other than catumaxomab, cancer, chemo- or radiotherapy
* previous treatment with entirely murine monoclonal antibodies other than catumaxomab
* liver metastases with volume >70 % of liver metastasized tissue

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-11; Primary Completion 2011-04 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
proportion of patients who are able to receive a second cycle of catumaxomab | 1 month

SECONDARY OUTCOMES:
puncture free survival | 1-3 months
incidence and severity of adverse events | 1 month
Quality of Life | 1 month
Development of human-anti-mouse antibodies | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Jalid Sehouli, MD, Prof, Principal Investigator — Charité Campus Virchow Clinic Berlin
Locations (1):
- Charité Campus Virchow Clinic, Berlin, Germany

REFERENCES:
- [Background] Heiss MM, Strohlein MA, Jager M, Kimmig R, Burges A, Schoberth A, Jauch KW, Schildberg FW, Lindhofer H. Immunotherapy of malignant ascites with trifunctional antibodies. Int J Cancer. 2005 Nov 10;117(3):435-43. doi: 10.1002/ijc.21165. PMID 15906359
- [Background] Ruf P, Lindhofer H. Induction of a long-lasting antitumor immunity by a trifunctional bispecific antibody. Blood. 2001 Oct 15;98(8):2526-34. doi: 10.1182/blood.v98.8.2526. PMID 11588051
- [Background] Riesenberg R, Buchner A, Pohla H, Lindhofer H. Lysis of prostate carcinoma cells by trifunctional bispecific antibodies (alpha EpCAM x alpha CD3). J Histochem Cytochem. 2001 Jul;49(7):911-7. doi: 10.1177/002215540104900711. PMID 11410615
- [Background] Zeidler R, Mysliwietz J, Csanady M, Walz A, Ziegler I, Schmitt B, Wollenberg B, Lindhofer H. The Fc-region of a new class of intact bispecific antibody mediates activation of accessory cells and NK cells and induces direct phagocytosis of tumour cells. Br J Cancer. 2000 Jul;83(2):261-6. doi: 10.1054/bjoc.2000.1237. PMID 10901380
- [Background] Zeidler R, Reisbach G, Wollenberg B, Lang S, Chaubal S, Schmitt B, Lindhofer H. Simultaneous activation of T cells and accessory cells by a new class of intact bispecific antibody results in efficient tumor cell killing. J Immunol. 1999 Aug 1;163(3):1246-52. PMID 10415020